CLINICAL TRIAL: NCT00405600
Title: A Prospective Randomized Clinical Investigation of Posterolateral Lumbosacral Spinal Fusions With BMP-2 and Titanium Pedicle Screw Instrumentation Versus BMP-2 Alone.
Brief Title: Spine Fusion Instrumented With BMP-2 vs Uninstrumented With Infuse BMP-2 Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, David Alexander, Principal Investigator, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA016
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Degenerative Lumbar Disc Disease; Spondylolisthesis; Spinal Stenosis
Keywords: Lumbar degenerative disease; spinal stenosis; spondylolisthesis; non instrumented surgery; instrumented surgery; BMP-2
MeSH Terms: conditions — Spondylolisthesis; Spinal Stenosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device (Active Comparator): Device used in surgery with or without instrumentation
  Interventions: Procedure: Device used in surgery with or without instrumentation

INTERVENTIONS:
Procedure: Device used in surgery with or without instrumentation — Infuse Bone Graft BMP-2, Large Kit will be used in all surgeries. Spine surgeries will be either instrumented or uninstrumented.

SUMMARY:
The goal of spinal fusion is to relieve pain and/or increase stability in painful or unstable spine joints. A patient may or may not receive rods and screws with the use of bone graft materials to facilitate bone growth and a fusion thus preventing movement of the bones of the spine.

In this research study, bone graft substitute material called Bone Morphogenetic Protein-2 known as BMP-2 Infuse will be used. No hip bone will be used. The surgical procedure will consist of BMP-2 Infuse with or without the use of rods and screws.

DETAILED DESCRIPTION:
In this study we will be using BMP-2 Infuse instead of the iliac crest bone graft for the spinal fusion. The BMP-2 Infuse has been researched in the only completed clinical trial for spinal fusions. It has demonstrated equivalence to the iliac crest bone graft with regard to both fusion rate and clinical outcome.

Currently, the acceptable standard of care for spinal fusion surgery requires instrumented or non-instrumented procedure with the use of bone graft materials, to facilitate bone growth, and a fusion, thus eliminating movement between the inciting vertebrae.

In this study, the surgical procedure will be BMP-2 Infuse with instrumentation or BMP-2 Infuse alone.

ELIGIBILITY:
Inclusion criteria:

* Patient not currently participating in a drug or medical clinical trial.
* Patient signed informed consent.
* Patient is willing to be available for each examination scheduled over the study duration.
* Patient has clinical and radiologic history of degenerative disc disease or spondylolisthesis (no greater than grade 1 utilizing Meyerding's classification (Meyerding HW, 1932)); spinal stenosis for which conservative treatment has failed and lumbar spinal fusion is indicated.
* Eligible for non-instrumented or instrumented surgical procedure
* Has one or two levels (contiguous) involvement from L1-S1 requiring fusion
* Has preoperative Oswestry score greater than 30
* Has not responded to non-operative treatment for a period of 6 months (bed rest, physical therapy, medication, manipulations, spinal injections, other).
* Is at least 20 years of age inclusive at the day of surgery
* If female of childbearing potential, patient is non-pregnant, non-nursing, and agrees to use adequate contraception for one year following surgery.

Exclusion Criteria:

* Patient has a systemic infection.
* Patient has had more than one previous non-fusion spinal surgery at the involved level.
* Patient requires fusion at more than 2 levels.
* Patient has pseudoarthroses from a previous fusion attempt.
* Patient has highly communicable diseases, inflammatory or autoimmune disease (e.g.osteomyelitis, crohn's, rheumatoid arthritis, systemic lupus, gout, HIV/AIDS, active tuberculosis, venereal disease, active hepatitis). A note to file written by the investigator will permit a patient into the study who experiences a mild case which will not affect the outcome of the study.
* Has been previously diagnosed with osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated
* Patient has a significant medical history that, in the Investigator's opinion would not make them a good study candidate.
* Patient requires interbody cage fusion or non-pedicle screw instrumentation.
* Pregnancy.
* Has presence of active malignancy (except basal cell carcinoma of the skin)
* Has a history of severe allergy (anaphylaxis)
* Is grossly obese, i.e. weight over 40% over ideal for their height and age.
* Has a fever (temperature over 101 F oral)
* Has an allergy to the BMP-2
* Has allergy to bovine products
* Has an allergy to collagen implants
* Is mentally incompetent(if questionable, obtain psychiatric consult)
* Is a prisoner, a transient or have been treated in an inpatient substance abuse program for alcohol and/or drug abuse within six months prior to proposed study enrollment.
* Has received drugs which may interfere with bone metabolism within two weeks prior to the planned surgery
* Has a diagnosis, which requires postoperative medication that interferes with fusion, such as steroids.
* Has history of endocrine or metabolic disorder known to affect osteogenesis (e.g. Paget's disease, renal osteodystrophy, Ehlers-Danios syndrome or osteogenesis imperfecta)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate bone fusion; | 3mon., 6mon., 12mon., 24mon
Radiology tests; CT spine 24mon. | 3mon., 6mon., 12mon., 24mon
Clinical neurological evaluations; patient questionnaires | 3mon., 6mon., 12mon., 24mon

SECONDARY OUTCOMES:
Hospital and surgical data | hospitalization;
Adverse events | hospitalization, clinic visits, unscheduled visits

CONTACTS AND LOCATIONS:
Overall Officials: Dr. David Alexander, M.D., Principal Investigator — Capital Health District Authority, Centre for Clinical Research, Queen Elizabeth II, Health Sciences Centre, 1278 Tower Rd.,Halifax, Nova Scotia, B3H-9Z9, Canada
Locations (1):
- Capital Health Health Authority, QEII Health Sciences Centre, Halifax Infirmary site,, Halifax, Nova Scotia, Canada